CLINICAL TRIAL: NCT06388785
Title: Post-vaccination Surveillance for Monitoring the Adverse Events Following Immunisation With QDENGA in a Real-world Setting in Malaysia (PRIME-Q)
Brief Title: A Study to Monitor the Adverse Events of QDENGA Vaccine in Participants in Malaysia
Acronym: PRIME-Q
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-003-5001
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Dengue Fever
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- QDENGA Vaccinated: Participants who have received QDENGA vaccine will be prospectively surveyed and regularly contacted to obtain data for up to 15 months post-vaccination.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The main aim of this study is to collect the number and type of medical problems (adverse events) after vaccination with QDENGA in Malaysia and to learn more about such medical problems after vaccination. Another aim of this study is to collect the number of persons vaccinated with QDENGA who need to stay in the hospital because of severe dengue fever.

No vaccination will be given as part of this study. The study will only collect data of persons already vaccinated with QDENGA who agree to participate.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have received at least one dose of QDENGA vaccine in Malaysia during the study period.
2. Participants or their legally authorized representative (LARs) with a functioning phone number.

Exclusion Criteria:

No exclusion criteria will be applied for this study.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants who have received the QDENGA vaccine in Malaysia and provided informed consent to participate in the active surveillance and data collection will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2027-05-08 (Estimated); Study Completion 2027-05-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From 14 days after first vaccination up to 15 months
  An AE is any untoward medical occurrence in a participant administered a studied drug and which does not necessarily have to have a causal relationship with the vaccine. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, a new disease or worsening in severity or frequency of a concomitant disease, temporally associated with the use of a studied drug, whether or not the event is considered causally related to the use of the product. An SAE is any untoward medical occurrence that at any dose: results in death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent, significant disability/incapacity, a congenital abnormality/birth defect, an important medical event in the opinion of the healthcare provider, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition above.

SECONDARY OUTCOMES:
Number of Participants who Require Hospitalization for Severe Dengue Diagnosed by Healthcare Provider (HCP) | From 14 days after first vaccination up to 15 months
  Number of participants who require hospitalization for severe dengue diagnosed by HCP will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Malaysia (2):
  - Universiti Malaya, Kuala Lumpur, Kuala Lumpur
  - Universiti Putra Malaysia, Serdang, Selangor

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link — https://clinicaltrials.takeda.com/study-detail/cbaebb4581e14b78??page=1&idFilter=TAK-003-5001